CLINICAL TRIAL: NCT04518813
Title: An Explorative Study of a Novel Non-invasive Glucose Measuring Device in Out-patient Settings
Brief Title: A Study of a Non-invasive Glucose Measuring Device in Out-patient Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RSP-24
Record Dates: First submitted 2020-08-13; First posted 2020-08-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus
Keywords: Non-invasive glucose monitoring; Raman spectroscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RSP-24 (Experimental): Subjects will perform calibrations on the IMD (Prototype 0.5) for 41 days over a 60 day period.
  Interventions: Device: Prototype 0.5

INTERVENTIONS:
Device: Prototype 0.5 — Investigational Medical Device collecting Raman data from tissue

SUMMARY:
This explorative clinical investigation has been launched to collect spectral Raman data paired with validated glucose reference values in persons with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects minimum 18 years of age
* Individuals diagnosed with any type of insulin-dependent diabetes mellitus ≥ 1 year
* Willing to perform up to 12 finger-pricks during each day of out-patient measurements
* Signed informed consent
* For women of childbearing potential: Willing and able to practice FDA approved birth control during the duration of the investigation
* Subject has a 2.4 GHz wireless internet connection at home (standard in normal routers) to be used in the study

Exclusion Criteria:

* For female subjects: Pregnancy or breastfeeding
* Skin phototype VI categorized by Fitzpatrick scale measured on thenar
* Subjects not able to understand and read local language
* Cognitive impairment, or in investigator's opinion, subject is not able to follow instructions provided and as specified in the protocol
* Subject not able to hold hand/arm steady (including tremors and Parkinson's Disease)
* Extensive skin changes, tattoos or diseases on right thenar (measurement site)
* Reduced circulation in right hand evaluated by Allen's test
* Known allergy to medical grade alcohol
* Hemodialysis
* Systemic or topical administration of glucocorticoids at the right hand for the past 7 days or during the study period expected
* Any disorder, which in the investigator's opinion might jeopardize subject's safety or compliance with the protocol
* Severe diabetes-related complications such as advanced autonomic neuropathy, kidney disease, foot ulcers, legal blindness, or symptomatic cardiovascular disease as evidenced by a history of cardiovascular episode(s)
* Dependency from the sponsor or the clinical investigator (e.g. co-workers of the sponsor, the study site, and/ or their families)
* Subjects currently participating in another study
* Subjects who have participated in the study IDT-1904-RO/RSP-21 or RSP-19.
* Incapacity for consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
Determination of number of calibration days | 2 years
  The number of calibration days needed for reaching a well-performing glucose predictive calibration model will be determined. The clinical performance of the reduced calibration model will be based on the data from the validation part by studying linear regression, Inter Subject Unified Performance value and Consensus Error Grid.
Safety evaluation of the Investigational Medical Device by reporting of adverse events | 2 years
  Safety of the IMD will be evaluated in a descriptive manner by the paucity of adverse events reported during the clinical investigation

SECONDARY OUTCOMES:
Device function | 2 years
  Device function will be evaluated in regard to durability and reliability. This is evaluated by reported device deficiencies during the study in the terms of subject diaries

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie, Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany